CLINICAL TRIAL: NCT04140968
Title: Impact of Progesterone Substitution in Luteal Phase on Resting Energy Expenditure in Women During Menopausal Transition.
Brief Title: Progesterone and Resting Energy Expenditure
Acronym: P4&REE
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: massive recruitment problems became apparent because of the strict inclusion criteria of our study.
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-01240
Record Dates: First submitted 2019-09-27; First posted 2019-10-28 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Menopause; Progesterone; Weight Gain
Keywords: Resting energy expenditure
MeSH Terms: conditions — Weight Gain | interventions — Utrogestan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Utrogestan (Experimental): 300mg Utrogestan (1 tablet 100mg + 1 tablet 200mg)by mouth,every day in the second and third menstrual cycle daily from cycle day 15 to 26.
  Interventions: Drug: Utrogestan

INTERVENTIONS:
Drug: Utrogestan — 300mg Utrogestan (1 tablet 100mg + 1 tablet 200mg) in the second and third menstrual cycle daily from cycle day 15 to 26.

SUMMARY:
This study evaluates the effect of micronized progesterone substitution in the luteal phase on resting energy expenditure in women during menopausal transition.

DETAILED DESCRIPTION:
The majority of women report an increase of body weight of about 0.5 kg/year during the menopausal transition. However, the weight gain has not been attributed to menopause itself but rather to, e.g., a decrease of the basal metabolic rate due to aging, less energy expenditure and a non-adapted caloric intake.

One of the first signs of the menopausal transition is a change in the bleeding pattern due to a disruption of the hypothalamus-pituitary-ovary-axis. The number of cycles with an insufficient luteal phase and anovulatory cycles with an insufficient or even absent luteal phase increase as the menopausal transition proceeds. Thus, in perimenopausal women progesterone endogenous exposure decreases in quantity and duration. By substituting progesterone during the luteal phase, irregular cycle and bleeding patterns can be normalized. However, besides the beneficial effects of progesterone on the course of a menstrual cycle it displays some features that may be preventive for weight gain.

In this study only women in their early menopausal transition with menstrual cycle irregularities are included. By substituting progesterone during luteal phase the investigator tries to normalize their menstrual cycle pattern. The hypothesis is, that progesterone might not only normalize the menstrual cycle pattern of women in their early menopausal transition but due to its metabolic activities, progesterone may also increase the resting energy expenditure and thus may prevent weight gain during the menopausal transition. Furthermore the effect of progesterone substitution on the expression of miRNAs which are included in glucose- and lipid-metabolism such as miR-370 and miR-29 will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Women during early menopausal transition (MT) with indication for luteal phase progesterone substitution (definition of early MT: change of cycle length (shorter or longer menstrual cycle) of at least ≥ 7 days from normal and/or phases of amenorrhea of up to < 60 days during the preceding 12 months)
* Body Mass Index (BMI) 18.5 - 24.9 kg/m2
* Informed Consent as documented by signature

Exclusion Criteria:

* Pregnancy or Lactation
* Systemic hormone therapy or hormonal contraception (estradiol, progestogen, androgen) during the study and within 12 weeks prior to study entry
* Phytotherapeutics for menstrual cycle regulation during the study and within 12 weeks prior to study entry
* Active psychiatric disease
* Use of psychotropic drugs during the study and within 12 weeks prior to study entry
* Nicotin abuse > 10 cigarettes/day
* Alcohol abuse
* Use of appetite suppressants
* Diabetes mellitus
* Untreated Hypo- and hyperthyroidism
* Hypersensitivity to progesterone
* Hypersensitivity to sunflower oil, soy lecithin and other ingredients of Utrogestan® such as gelatine, glycerol, E171 (titanium dioxide)
* Contraindication of progesterone medication according to swissmedicinfo.ch (suspected or diagnosed neoplasia of the breast or other sexual organ; benign or malignant liver Tumors (also in medical history); acute or chronic liver disease (Rotor- or Dubin-Johnson-Syndrome); cholestatic jaundice; porphyria; arterial or venous thromboembolic Events and cerebral bleedings; abnormal genital bleeding of unknown cause)
* Use of barbiturates, antiepileptic drugs, tuberculostatic drugs, antiretroviral drugs, antimycotic drugs, antibiotic drugs, Hypericum perforatum and Spironolactone
* Known or suspected non-compliance, drug or alcohol abuse etc.
* Illiteracy
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 2 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-05-27 (Actual); Study Completion 2021-05-27 (Actual)

PRIMARY OUTCOMES:
Mean change in resting energy expenditure | cycle 1 (day 20) to cycle 3 (day 20), (cycle 1 has individual length, <60 days, cycle 2&3 are 28 days)
  Change in resting energy expenditure (kcal/day) from cycle 1 due to substitution of Utrogestan in luteal phase

SECONDARY OUTCOMES:
Mean change in miRNA expression | cycle 1 (day 5; day 20) and cycle 3 (day 5; day 20), (cycle 1 has individual length, <60 days, cycle 2&3 are 28 days)
  Change in miRNA expression (miR-370, miR-29b)
Mean change in energy intake | cycle 1 (day 17-19) and cycle 3 (day 17-19), (cycle 1 has individual length, <60 days, cycle 2&3 are 28 days)
  Change in energy intake (kcal/day)
Mean change in body core temperature | cycle 1-3 during luteal phase, (cycle 1 has individual length, <60 days, cycle 2&3 are 28 days)
  Change in body core temperature (°C)
Mean change in serum hormone profile FSH | cycle 1 (day 5; day 20) and cycle 3 (day 5; day 20), (cycle 1 has individual length, <60 days, cycle 2&3 are 28 days)
  Change in serum hormone profile: FSH (U/l)
Mean change in serum hormone profile LH | cycle 1 (day 5; day 20) and cycle 3 (day 5; day 20), (cycle 1 has individual length, <60 days, cycle 2&3 are 28 days)
  Change in serum hormone profile: LH (U/l)
Mean change in serum hormone profile estradiol | cycle 1 (day 5; day 20) and cycle 3 (day 5; day 20)
  Change in serum hormone profile: estradiol (pmol/l)
Mean change in serum hormone profile progesterone | cycle 1 (day 5; day 20) and cycle 3 (day 5; day 20), (cycle 1 has individual length, <60 days, cycle 2&3 are 28 days)
  Change in serum hormone profile: progesterone (nmol/l)
Mean change in fasting glucose | cycle 1 (day 5; day 20) and cycle 3 (day 5; day 20), (cycle 1 has individual length, <60 days, cycle 2&3 are 28 days)
  Change in fasting glucose (mmol/l)
Mean change in fasting Insulin | cycle 1 (day 5; day 20) and cycle 3 (day 5; day 20), (cycle 1 has individual length, <60 days, cycle 2&3 are 28 days)
  Change in fasting Insulin (mU/l)
Mean change in blood lipid serum level: cholesterol | cycle 1 (day 5; day 20) and cycle 3 (day 5; day 20), (cycle 1 has individual length, <60 days, cycle 2&3 are 28 days)
  Change in cholesterol (mmol/l)
Mean change in blood lipid serum level: LDL | cycle 1 (day 5; day 20) and cycle 3 (day 5; day 20), (cycle 1 has individual length, <60 days, cycle 2&3 are 28 days)
  Change in LDL (mmol/l)
Mean change in blood lipid serum level: HDL | cycle 1 (day 5; day 20) and cycle 3 (day 5; day 20), (cycle 1 has individual length, <60 days, cycle 2&3 are 28 days)
  Change in HDL (mmol/l)
Mean change in blood lipid serum level: triglycerides | cycle 1 (day 5; day 20) and cycle 3 (day 5; day 20), (cycle 1 has individual length, <60 days, cycle 2&3 are 28 days)
  Change in triglycerides (mmol/l)

CONTACTS AND LOCATIONS:
Overall Officials: Petra Stute, Prof, Principal Investigator — University Hospital Berne
Locations (1):
- Dep. of Obstetrics and Gynecology, Bern University Hospital, Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No